CLINICAL TRIAL: NCT02124330
Title: Protein Sorbent Properties of Montmorillonite in Vitro and in Vivo Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luca Ronfani (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor-Investigator, Luca Ronfani, Dr, IRCCS Burlo Garofolo
Organization: IRCCS Burlo Garofolo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 06-13; RC 06/13 (Other: IRCCS Burlo Garofolo)
Record Dates: First submitted 2013-10-21; First posted 2014-04-28 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Urea Cycle Disorders, Inborn; Other Metabolic Diseases
Keywords: Montmorillonite, proteic diet, in vitro and in vivo models
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — Bentonite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- montmorillonite 5 g (Experimental): 5g Montmorillonite + 15 g protein (ratio 1:3)
  Interventions: Dietary Supplement: montmorillonite 5 g
- Montmorillonite 3 g (Experimental): 3g Montmorillonite + 15 g protein (ratio 1:5)
  Interventions: Dietary Supplement: montmorillonite 3 g
- Montmorillonite 1 g (Experimental): 1g Montmorillonite + 15 g protein (ratio 1:15)
  Interventions: Dietary Supplement: Montmorillonite 1 g
- Control (No Intervention): A control goup will intake 15 g of protein alone

INTERVENTIONS:
Dietary Supplement: montmorillonite 5 g — 5g montmorillonite + 15 g protein (ratio 1:3)
  Arms: montmorillonite 5 g
Dietary Supplement: montmorillonite 3 g — 3g MONT+ 15 g protein (ratio 1:5)
  Arms: Montmorillonite 3 g
Dietary Supplement: Montmorillonite 1 g — 1g MONT+ 15 g protein (ratio 1:15)
  Arms: Montmorillonite 1 g

SUMMARY:
Montmorillonite (MONT) is a phyllosilicate layered mineral with unique physicochemical properties, such as swelling and cation exchange capability.

The aim of this project is to study, in healthy volunteers, the in vivo ability of MONT to reduce protein intestinal uptake. Furthermore, the study analyzed in vitro the MONT ability of immobilizing proteins.

DETAILED DESCRIPTION:
Montmorillonite (MONT) is a phyllosilicate layered mineral; chemically it is hydrated sodium calcium aluminium magnesium silicate hydroxide. Potassium, iron, and other cations are common substitutes and the exact ratio of cations varies with source.

Due to its unique physicochemical properties, such as swelling and cation exchange capability, as well its mechanical and thermal stability, MONT can be efficiently used as matrix for immobilization of proteins with high molecular weight (e.g. Albumin) and proteins with low molecular weight (e.g.Aflatoxines). Therefore, MONT is used for therapeutic purposes, in pharmaceutical formulations and in food preparations. In vitro assays made in our laboratory, showed that MONT absorbs, in stable manner, alimentary proteins: beta-lactoglobulins, alfa lactoalbumines and the ratio MONT-protein (w/w) 1:3, 1:5, 1:15, results in the protein capture of 50, 27, 0 % of proteins respectively.

The aim of this project is to study, in healthy volunteers, the in vivo ability of MONT to reduce protein intestinal uptake evaluated with the blood MONT- protein ratio. Furthermore, the study analyzed in vitro the MONT ability of immobilizing proteins at different ratio (w/w) 1:3, 1:5, 1:15.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (12M, 13 F, 25-30 years). Fasting from morning

Exclusion Criteria:

* not defined

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Protein uptake evaluated with the blood MONT-protein ratio | before administration and 30, 60, 90, 120 ,180 minutes after
  A solution of MONT and whey protein dissolved in 200 ml of water at the three different ratios will be administered. The control group will intake 15g of protein alone.
  Blood samples will be centrifuged and analyzed by mass spectrometry (egilent HP5973 mass spectrometry).

SECONDARY OUTCOMES:
Protein absorption by MONT in vitro | at time of the trial
  MONT and protein (whey protein) at three different ratio w/w (1:3, 1:5, 1:15) will be dissolved in acetate buffer 0.1M pH5 as well as a sample without MONT.
  Samples will incubate at RT for 1, 10, 30, 60 minutes and then centrifugate at 13000g.
  The surnatant will be analyzed by LOWRY method. Protein concentration will be expressed in mg/ml. The MONT ability of immobilization will be calculated respect to the protein control sample

CONTACTS AND LOCATIONS:
Overall Officials: Tarcisio Not, MD, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy